CLINICAL TRIAL: NCT00855075
Title: Correlation of the Cerebral State Index With the Richmond Agitation-Sedation Scale in ICU Patients Who Are Sedated and Mechanically Ventilated: A Pilot Study
Brief Title: Correlation of Cerebral State Index With the Richmond Agitation-Sedation Scale in Mechanically Ventilated ICU Patients
Status: Terminated | Type: Observational
Why Stopped: Technology used to obtain/measure cerebral state index is no longer manufactured
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Audis Bethea, Pharm.D., Clinical Pharmacy Specialist, CAMC Health System
Other Study IDs: 08-03-2038
Record Dates: First submitted 2009-01-15; First posted 2009-03-04 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sedation; Analgesia
Keywords: Sedation; Analgesia; Mechanical ventilation; Cerebral State Monitor; Cerebral State Index
MeSH Terms: conditions — Agnosia | interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral State Monitor: A cerebral state monitor will provide a cerebral state index for mechanically ventilated intensive care patients. Recorded cerebral state indexes will be correlated with clinical assessments of sedation using the Richmond Agitation-Sedation Scale.
  Interventions: Device: Cerebral State Monitor

INTERVENTIONS:
Device: Cerebral State Monitor — A cerebral state monitor will provide a cerebral state index for mechanically ventilated intensive care patients. Recorded cerebral state indexes will be correlated with clinical assessments of sedation using the Richmond Agitation-Sedation Scale.
  Other Names: Danmeter; Cerebral State Index

SUMMARY:
The purpose of this study is to correlate the cerebral state index obtained from a cerebral state monitor with the Richmond Agitation-Sedation Scale assessment performed on sedated and mechanically ventilated intensive care patients.

DETAILED DESCRIPTION:
Currently there are no objective methods to measure levels of sedation in all ICU patient populations. This generally does not become problematic in most patients. However, certain populations cannot be assessed by standard means. These populations would include patients who are quadriplegic and those who are being treated with neuromuscular blocking agents. The current norm is to use a sedation scale such as the Richmond Agitation-Sedation Scale to assess the patient's level of sedation. An alternative to this would be to use an EEG based method that monitors brain activity. New methods of monitoring brain activity, using cerebral state monitors may provide an effective means of monitoring sedation. The cerebral state monitor, however, and the parameters it provides, the cerebral state index, has not been tested in an ICU setting. Correlating the measurements gained from the cerebral state monitor with the RASS assessment from sedated ICU patients may allow us to develop a method of monitoring sedation in populations that were impossible to monitor previously. Accurately monitoring the level of sedation in these patients may help decrease the incidence of over-sedation and under-sedation.

ELIGIBILITY:
Inclusion Criteria:

* Admission the surgical-trauma intensive care unit at the Charleston Area Medical Center General Hospital
* Adult (18-85 years of age)
* Anticipated duration of mechanical ventilation of at least 72 hours

Exclusion Criteria:

* Patients admitted with paralysis or a brain injury
* Patients who are deaf, blind, or have pre-existing dementia/delirium

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults admitted to the surgical-trauma unit at Charleston Area Medical Center with an anticipated duration of mechanical ventilation of at least 72 hours.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Correlation of cerebral state index and Richmond Agitation-Sedation Scale | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Audis Bethea, PharmD, BCPS, Principal Investigator — Charleston Area Medical Center Health System
Locations (2):
- United States (2):
  - Charleston Area Medical Center, General Hospital, Charleston, West Virginia
  - Charleston Area Medical Center Health System, Charleston, West Virginia

REFERENCES:
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Jensen EW, Litvan H, Revuelta M, Rodriguez BE, Caminal P, Martinez P, Vereecke H, Struys MM. Cerebral state index during propofol anesthesia: a comparison with the bispectral index and the A-line ARX index. Anesthesiology. 2006 Jul;105(1):28-36. doi: 10.1097/00000542-200607000-00009. PMID 16809991
- [Background] Zhong T, Guo QL, Pang YD, Peng LF, Li CL. Comparative evaluation of the cerebral state index and the bispectral index during target-controlled infusion of propofol. Br J Anaesth. 2005 Dec;95(6):798-802. doi: 10.1093/bja/aei253. Epub 2005 Oct 6. PMID 16210310
- [Background] Anderson RE, Jakobsson JG. Cerebral state monitor, a new small handheld EEG monitor for determining depth of anaesthesia: a clinical comparison with the bispectral index during day-surgery. Eur J Anaesthesiol. 2006 Mar;23(3):208-12. doi: 10.1017/S0265021505002206. PMID 16430792
- [Background] Hernandez-Gancedo C, Pestana D, Perez-Chrzanowska H, Martinez-Casanova E, Criado A. Comparing Entropy and the Bispectral index with the Ramsay score in sedated ICU patients. J Clin Monit Comput. 2007 Oct;21(5):295-302. doi: 10.1007/s10877-007-9087-7. Epub 2007 Aug 16. PMID 17701384
- [Background] Sydow M, Neumann P. Sedation for the critically ill. Intensive Care Med. 1999 Jun;25(6):634-6. doi: 10.1007/s001340050917. No abstract available. PMID 10416920
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Vereecke HE, Vanluchene AL, Mortier EP, Everaert K, Struys MM. The effects of ketamine and rocuronium on the A-Line auditory evoked potential index, Bispectral Index, and spectral entropy monitor during steady state propofol and remifentanil anesthesia. Anesthesiology. 2006 Dec;105(6):1122-34. doi: 10.1097/00000542-200612000-00012. PMID 17122575